CLINICAL TRIAL: NCT06190106
Title: Experiences of Psychotherapeutic Outcomes in Women Victims of Domestic Violence
Acronym: EPOWVDV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Government College University Faisalabad (Other)
Responsible Party: Principal Investigator, Qasir Abbas, Dr. Qaisir Abbas Assisstant Professor Clinical Psychology, Government College University Faisalabad
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: GovernmentGCUF
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Experiences of Psychitherapeutic Outcomes in Women Victims of Domestic Violence
Keywords: Domestic Violence, Psychotherapy, Psychiatric Symptoms, Intimate Partner Victimization (IPV)
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: only a single group is studied and their experiences are explored first after screening the psychiatric symptoms of depression, anxiety, and stress and then providing them with Cognitive Behavioral interventions to check the improvement in their Psychiatric symptoms and assess the positive and negative aspects and outcomes of Psychotherapeutic Intervention,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental treatment group (Experimental): Participants had received 8-10 cognitive behavior therapy-based therapeutic sessions and their feedback was taken to check the positive and negative effects of Psychotherapeutic Intervention (cognitive-behavioral intervention).
  Interventions: Other: Cognitive Behavioral Therapy (Psychotherapeutic Intervention)

INTERVENTIONS:
Other: Cognitive Behavioral Therapy (Psychotherapeutic Intervention) — A psychotherapeutic intervention CBT is given to assess the improvement and betterment in mental health and to assess the reduction of Psychiatric symptoms like depression, anxiety and stress

SUMMARY:
The main objectives of the study are:

1. To explore the experience of undergoing psychotherapy of women victims of domestic violence.
2. To explore the effects of undergoing psychotherapy among women with victims of domestic violence.

DETAILED DESCRIPTION:
Participants:

Purposive sampling techniques would be followed to inquire about the data from the sample. The sample of the present study would be the women who are victims of domestic violence. The study's sample size is 15 which pre and post-testing would be implied. The participants were briefed about the objectives of the present study. Informed consent was taken to ensure the willingness of the participants. First, the DASS test is fulfilled to check out the symptoms caused by domestic violence in women. To fulfill the criteria, they inquired about the topic in detail to get in-depth information from the participants about their experiences and mental health problems caused by domestic violence. Later, they were provided with psychotherapeutic sessions to treat or reduce their mental health problems, and again an in-depth interview about these therapy sessions was conducted to check the effectiveness of the treatment given.

ELIGIBILITY:
Inclusion Criteria:

* the participants that would be included in the study are females who would be victims of Domestic Violence with the age range of 18 years to 45 years and women who would be eligible for taking psychotherapeutic intervention

Exclusion Criteria:

* women with psychotic disorders would be excluded and those who wouldn't meet the criteria of the DASS test

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — only women who are the victims of domestic violence and who fulfilled the criteria of DASS and then taken Cognitive-behavioral Interventions.
Enrollment: 15 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-04-10 (Estimated)

PRIMARY OUTCOMES:
Depression anxiety and stress scale | 4 months
  Depression anxiety and stress scale would be used at pre-assessment and post-assessment stage to investigate the impact of ongoing psychotherapy, using qualitative interviews

CONTACTS AND LOCATIONS:
Overall Officials: Qasir Abbas, PHD, Principal Investigator — Government College University Faisalabad
Locations (1):
- Department of Applied Psychology, Faisalābad, Pakistan

IPD SHARING:
Plan to Share IPD: No